CLINICAL TRIAL: NCT04211740
Title: Efficacy and Safety of OCH-NCNP1 in Patients With Relapsing Multiple Sclerosis
Brief Title: Phase II Clinical Trial of OCH-NCNP1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Principal Investigator, Tomoko Okamoto, Medical director, National Center of Neurology and Psychiatry, Japan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCH-NCNP1-02
Record Dates: First submitted 2019-12-17; First posted 2019-12-26 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCH-NCNP1 3 mg (Active Comparator)
  Interventions: Drug: OCH-NCNP1
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OCH-NCNP1 — OCH-NCNP1 3mg is supplied as granules and take orally once a week.
  Arms: OCH-NCNP1 3 mg
Drug: Placebo — Placebo is supplied as granules and take orally once a week.
  Arms: Placebo

SUMMARY:
This study is designed to assess the efficacy and safety of OCH-NCNP1 compared to placebo in subjects diagnosed with relapsing remitting multiple sclerosis (RRMS) and secondary progressive mltiple sclerosis (SPMS) .

ELIGIBILITY:
Inclusion Criteria:

* Subject with Multiple Sclerosis eligible for enrolment in the study must meet all of the following criteria:

  1. Provision of written informed consent to participate in this study
  2. Patients diagnosed as relapsing remitting multiple sclerosis based on modified McDonald criteria in 2017
  3. Relape must have been confirmed by a neurologist at least twice within 24 months, or once within 12 months before enrollment
  4. Have at least one T2 lesion on MRI scans at screening
  5. EDSS less than or equal to 7
  6. 20 =< Age < 65
  7. Promise to prevent conception for at least 90 days after the last administration
  8. Neurological stability has been confirmed by a neurologist

Exclusion Criteria:

* Subject with MS patients meeting any of the following criteria must not be enrolled in the study:

  1. Diagnosed as Neuromyelitis Optica
  2. Women who are pregnant or lactating
  3. Patients who is prohibited MRI
  4. Patients who are allergic to Gd-contrast medium
  5. History of liver diseases or liver transplantation
  6. Liver dysfunction in the screening test and baseline physical examination
  7. History of cancer past five years
  8. Negative for herpes zoster virus antibody
  9. Positive for Syphilis serum reaction
  10. Positive for Beta-glucan or positive for T-spot
  11. Positive for Anti-Aquaporin 4 antibody
  12. History of HIV infection
  13. History of HBV or HCV infection
  14. History of Transplantation
  15. Use of any other investigational agents and/or experimental agents within 4 months prior to the first anticipated administration of study medication.
  16. History of blood donation (200 ml within 2 months, 400 ml within 3 months) prior to the first anticipated administration of study medication
  17. Lymphocyte number < 600 /mm3 in peripheral blood
  18. Current diagnosed or suspected infectious diseases
  19. Compromised Patients
  20. Inflammatory Bowel disease
  21. Subjects with prolongation of QT/QTc interval
  22. History or have risk of torsade de pointes
  23. Taking the medicine which has risk of prolongation of QT/QTc interval
  24. History of severe allergy of medicine or food
  25. History or current of drug/ alcohol addiction
  26. Bronchial Asthma
  27. Epilepsy Other protocol-defined exclusion criteria may apply

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The rate of the patients who identified new or enlarging T2 lesions on MRI scans compared to baseline | Change from screening at Month 6.

SECONDARY OUTCOMES:
annual relapse rate | Month 6
Detection of asymptomatic | Month 6
Expanded Disability Status Scale (EDSS) / Functional Scale (FS) | screening, 4weeks, 8 weeks, 12 weeks, 16weeks, 20 weeks, 24 weeks
Duration of sustained reduction in disability (SRD) | Month 6
Change of MRI | Change from screening at Month 3 and 6
Change of No evidence of disease activity (NEDA) | Change from screening at Month 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Okamoto, MD, Principal Investigator — National Center of Neurology and Psychiatry
Locations (1):
- National Center of Neurology and Psychiatry, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okamoto T, Ishizuka T, Shimizu R, Asahina Y, Nakamura H, Shimizu Y, Nishida Y, Yokota T, Lin Y, Sato W, Yamamura T. Efficacy and Safety of the Natural Killer T Cell-Stimulatory Glycolipid OCH-NCNP1 for Patients With Relapsing Multiple Sclerosis: Protocol for a Randomized Placebo-Controlled Clinical Trial. JMIR Res Protoc. 2024 Jan 15;13:e46709. doi: 10.2196/46709. PMID 38224478